CLINICAL TRIAL: NCT05319041
Title: Randomised Placebo Controlled Study of Herbal Medication to Treat Dry Eye in Peri/ Post-menopausal Women
Brief Title: Herbal Medication to Treat Dry Eye in Peri/ Post-menopausal Women
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: Singapore Chung Hwa Medical Institution (Other)
Responsible Party: Principal Investigator, Louis Tong, Principal Investigator, Singapore National Eye Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R1675/72/2019; 2019/2957 (Other: SingHealth Centralised Institutional Review Board)
Record Dates: First submitted 2022-03-22; First posted 2022-04-08 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Dry Eye
Keywords: Menopausal women; Herbal treatment; Quality of Life; eicosanoids; cytokines
MeSH Terms: conditions — Dry Eye Syndromes | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active herbal capsules (Experimental): Wei's Qi Ju Gan Lu Formula is a herbal formulation initiated by the senior TCM collaborator, Prof Wei QP. This TCM formulation is prescribed to treat the dry eye patients with "liver-kidney yin deficiency". The treatment regulation aims to nourish the Liver and Kidney, enrich yin deficiency, in order to promote tears production, hence treatment of Dry Eye.
  Interventions: Drug: Wei's Qi Ju Gan Lu Formula
- Placebo capsules (Placebo Comparator): Placebo capsule which contains 0.5g maltodextrin without any herbs medicine.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Wei's Qi Ju Gan Lu Formula — The formulation, Wei's Qi Ju Gan Lu Formula, is initiated by the senior TCM collaborator, Prof Wei QP, is formulated to treat the dry eye patients with "liver-kidney yin deficiency". The treatment regulation aims to nourish the Liver and Kidney, enrich yin deficiency, in order to promote tears production, hence treatment of Dry Eye.
  Arms: Active herbal capsules
Drug: Placebo — 0.5g maltodextrin without any herbs medicine
  Other Names: 0.5g maltodextrin without any herbs medicine
  Arms: Placebo capsules

SUMMARY:
Dry eye disease (DED) in less severe forms are very common, and should ideally be treated outside hospitals, eg., through primary care services and exploiting holistic therapies such as traditional medicine. This will keep the care affordable and accessible despite a large burden of care.

Postmenopausal women, compared to others in the population, have a higher incidence of DED. Large-scale epidemiological studies done in the United States have shown that the rate of DED in women over 50 years old is nearly double that in men over 50, at 7% and 4%, respectively. Studies have demonstrated that there is a hormonal etiology behind this group's susceptibility to DED, although the precise hormonal imbalance and mechanistic pathway for DED are still unclear.

A significant number of women seen at the dry eye clinic are post-menopausal, and very symptomatic, though many do not have the corneal epitheliopathy evidenced by dye staining. Such patients are not likely to benefit from conventional prescription drugs for dry eye, such as cyclosporine and corticosteroids. Hormonal replacement therapy for menopausal women has not been universally accepted, and there may be an increased risk of carcinomas, on the other hand, topical hormonal therapy for dry eye is not widely available, and still controversial, so there is a definite unmet need for new therapeutic modalities to treat dry eye in post-menopausal women.

Traditional Chinese Medicine (TCM) is a form of complementary medicine that aims to treat yin or yang deficiency syndromes, using modalities like herbs, acupuncture or moxibustion. Menopause in women, particularly in Asia, has been linked to yin-deficiency, in one study, 73% of Chinese post-menopausal women suffered from kidney yin-deficiency. A review of randomized controlled trials of TCM treatment showed that certain modalities like soy and phytoestrogens have been useful in the treatment of syndromes in menopause, such as hot flushes.

DETAILED DESCRIPTION:
The overall hypothesis is that the Traditional Chinese Medicine (TCM) modality of a specific herbal formulation can improve the symptoms and signs of post-menopausal dry eye in women, and objectively, these improvements are associated with improvement of dry eye symptoms, and alteration of levels of tear eicosanoids or cytokines.

TCM in the treatment of dry eye A meta-analysis of TCM in treatment of Sjogren's syndrome showed that TCM is promising but there were some flaws in the studies reviewed.

Jiang et al, in particular has found that mistletoe, in combination with carboxymethylcellulose eyedrops were effective in reducing dry eye symptoms and signs, compared to normal saline eyedrops, in post-menopausal women.Unfortunately, the authors did not compare the effect of this combination with carboxymetholycellulose eyedrops, a commonly used artificial tear, per se.

In postmenopausal women, dry eye is not only more common, but the symptoms may be confused/related to mood changes like depression and anxiety, and sleep disorders, all of which were linked to the post-menopausal state, where there may be yin deficiency.

Recently the investigators found acupuncture to be useful in the treatment of elderly people with lung-kidney yin-deficiency type of dry eye in Singapore. In addition, TCM Practitioners in Singapore were interested in the treatment of dry eye. However, no study has evaluated the use of TCM herbs in peri-menopausal patients with dry eye in robust way.

Previous studies by the senior TCM collaborator, Prof Wei QP has concluded that steaming treatment by (Wei's Qi Ju Gan Lu Formula) combined with sodium hyaluronate eye drops could improve the objective indexes like TBUT and corneal staining as well as subjective symptoms in peri-menopausal patients with aqueous tear deficiency dry eye of liver and kidney deficiency. Prof Wei has also studied treatment of dry eye through oral medication (with the method of strengthening the water element to nourish wood element under the TCM perspective) combined with artificial tears, and concluded that the prescription can effectively treat dry eyes by promoting the tear secretion and prolonging BUT. Recently, the investigators have also discovered that herbal medication have a trend to lower the tear levels of inflammatory proteins (journal under review). Hence, this current study intends to follow-up with the effectiveness of oral medication of (Wei's Qi Ju Gan Lu Formula) for patients suffering from peri/ post-menopausal dry eye disease of the "Liver-Kidney yin deficiency" pattern differentiation.

1.1.1 Rationale for the Study Purpose Clinical significance Traditional Chinese Medicine (TCM), when combined with psychotherapy, has been shown to be effective in targeting yin-deficiency in the treatment of menopause, although the effect of such treatment on dry eye symptoms has not been specifically investigated.

If TCM is effective in the treatment of post-menopausal women, it can be implemented at the primary care level, so relieving the specialist centers of this type of patients, thereby saving health-care costs.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-79 years old women
2. Peri and Post-menopausal women
3. Chief complaint of participant should be consistent with dry eye symptoms based on SPEED Questionnaire, with a score of > 6 (Appendix 5)
4. History of presenting TCM score symptoms:

   4.1. TCM dry eye assessment score (Appendix 3) The pattern deviation can be determined if 3 or more main symptoms are present (one of which is a localized eye symptom and one of which is a system symptom), together with at least one accompanying symptom.

   4.2 Liver-Kidney yin deficiency assessment score (Appendix 4) This form is to determine the extent of Liver-Kidney Yin Deficiency (assessed at SCHMI).

   Any score<14 will not satisfy the criterion for Liver Kidney Yin Deficiency and will not be recruited. This detailed TCM score will also be a secondary outcome measure in the analysis of pre/post herbal treatment (see below).
5. Clinical signs:

   5.1. Tear break up time (TBUT) ≤10s or Schirmer I test ≤10mm/5 mins
6. Normal renal and liver function at baseline, i.e., all parameters within the reference value

Exclusion Criteria:

1. Currently or intention to use hormonal therapy (eg. cancer patients who is on tamoxifen)
2. Currently pregnant or breastfeeding
3. Hysterectomy procedure done previously
4. Removal of cysts or polyp procedure done previously
5. Requirement to wear contact lens, and having worn such lenses in week preceding eligibility
6. Glaucoma, significant cataract, age related macular degeneration or other ophthalmic disease, eg. Extraocular muscle palsies, facial paralysis, ectropion, entropion, trichiasis
7. Requirement of any eyedrops other than artificial tears.
8. Previous eye surgeries including LASIK (within 6 months) or punctal plugs in-situ
9. Autoimmune systemic diseases: Steven-Johnson syndrome, Sjogren's syndrome, Rheumatoid Arthritis, Lupus
10. Systemic disease requiring regular medication (except hypertension and lipidemia)

Ages: 40 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Peri and Post-menopausal women age between 40-79 years old
Enrollment: 150 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Change in SPEED score | 3 months
  To assess the improvement of dry eye symptoms by SPEED questionnaire. 0 score is the minimum (no dry eye symptom); 64 is the maximum score (most symptomatic)

SECONDARY OUTCOMES:
Change in SPEED score | 4 months
  To assess the improvement of dry eye symptoms by SPEED questionnaire. 0 score is the minimum (no dry eye symptom); 64 is the maximum score (most symptomatic)
Change in Sleep score | 3 months
  To assess the improvement of sleep score. 0 score is the minimum (no sleeping issue); 24 score is the maximum (high risk of Epworth Sleepiness Scale)
Change in Depression score | 3 months
  To assess the improvement in depression score. 0 score is the minimum (no sign of depression); 48 score is the maximum (very likely to have depression)
Change in TCM score (Liver-Kidney Yin Deficiency) | 3 months
  To assess the change in TCM score. Liver-Kidney Yin deficiency is within the range from 14-30. (score <14 not diagnosed as Liver-Kidney Yin Deficiency); (score 14-20 Liver-Kidney Yin deficiency Type I- Level 1 mild); (score 21-30 Liver-Kidney Yin deficiency Type II- Level 2 moderate); (score >30 Liver-Kidney Yin deficiency Type III- Level 3 severe)

CONTACTS AND LOCATIONS:
Overall Officials: Louis Tong, PhD, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No